CLINICAL TRIAL: NCT04540471
Title: Department of Nursing, Chang Gang Memorial Hospital
Brief Title: Music Therapy in Patients With Breast Cancer- a Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: miss contact
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201901698B0
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-01

CONDITIONS: Music Therapy, Breast Cancer, Anxiety, Fatigue
MeSH Terms: conditions — Breast Neoplasms; Anxiety Disorders; Fatigue | interventions — Music Therapy; Educational Status

STUDY DESIGN:
Intervention Model Description: an assessor blinded, randomized, controlled, parallel group trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Block randomisation was implemented (block size = 4). A random number generator was used to generate random numbers, and all participants were subsequently given an MP3 player.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT group (Experimental): The participants in MT group will receive music therapy 1 day per week for 1 hour with total 12hours in12 consecutive weeks after initial enrollment. Initial evaluation at the first session, including patient's vital sign, consciousness and spirit. The music therapy will consist of therapeutic singing, interpersonal communication, melody intonation therapy and rhythmic hands slapping. During therapeutic singing session, the music therapists will sing a song first and then the patients sing it after them. Interpersonal communication activity will be led by the music therapist and passed on to one patient to another patient. Melody intonation therapy will comprise communication, chatting and read aloud by using melody.
  Interventions: Other: music; Other: comprehensive in-patient education program
- Control group (Placebo Comparator): control groups will receive comprehensive in-patient education program for 12 consecutive weeks
  Interventions: Other: comprehensive in-patient education program

INTERVENTIONS:
Other: music — MT group receives additional music therapy
  Other Names: education
  Arms: MT group
Other: comprehensive in-patient education program — comprehensive in-patient education program

SUMMARY:
Comprehensive inpatient rehabilitation for breast cancer consist of interdisciplinary team care but few researchers investigate the efficacy of music therapy, which have shown some benefits in breast cancer rehabilitation. According to previous research, music therapy has been proposed to improve quality of life, as well as depression and stress of breast cancer patients. However, to the best of our knowledge, only few studies have investigated the impact of music therapy among health-related parameter of patient with breast cancer. Considering the fact that music therapy had merely no adverse events, we assume music therapy is an optimal add-on therapy for patient with breast cancer. Therefore, we plan to conduct a study to evaluate the impact of music therapy on anxiety, and fatigue on patients with breast cancer.

DETAILED DESCRIPTION:
Patients and Method:

We designed this study as an assessor blinded, randomized, controlled, parallel group trial. The participants will be recruited from general surgery unit of tertiary referral hospital in Southern Taiwan. Inclusion criteria will be as follows: (1) patients with first-ever breast cancer between 20~80 years old (1 to 6 months post- surgery) (2) able to follow basic orders (verbal or gesture) and tolerated music therapy by 1 hour. Individuals will be excluded from the study if they (1) are unable to cooperate with music therapy, (2) undergoing psychotherapeutic treatment during the study period, using antidepressants during the study period, (3) are significantly hearing impaired, not agree to sign the informed consent, or do not agree further evaluation, and (4) pregnant women. Randomization in a 1:1 ratio will be performed with computer-generated randomization list. All the included patients will be categorized into two groups: music therapy (MT) group and control group. Both groups will receive comprehensive in-patient education program for 12consecutive weeks, but the MT group will receive additional music therapy in the 12 consecutive weeks. The participants in MT group will receive neurologic music therapy 1 day per week for 1 hour with total 4 hours in 4 consecutive weeks after initial enrollment. The primary outcome is anxiety and fatigue. The Brief Fatigue Inventory-Taiwan (BFI-T) State anxiety inventory (STAI) and WHOQOL until 12 weeks after randomization. All health-related parameters will be evaluation prior to intervention and after intervention.

Aim of the study:

The aim of the study is to explore the impact of music therapy on anxiety and fatigue among patients with breast cancer. We aim to investigate whether music therapy is an optimal add-on therapeutic model for patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

- We design this study as an assessor blinded, randomized, controlled, parallel group trial. The participants will be recruited from OPD unit of tertiary referral hospital in Southern Taiwan. Inclusion criteria will be as follows: (1) patients with breast cancer between 20~80 years old at stage (1-6 months post surgery) (2) able to follow basic orders (verbal or gesture) and tolerated music therapy by 1 hour.

Exclusion Criteria:

Individuals will be excluded from the study if they are unable to cooperate with music therapy, are significantly hearing impaired, are severely mentally impaired (MMSE<10), or not agree to sign the informed consent, uncontrolled seizure or do not agree further evaluation. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
State anxiety inventory (STAI) Survey | 12 weeks
  We accessed anxiety by State anxiety inventory (STAI) it has 20 items for assessing trait anxiety and 20 for state anxiety. State anxiety items include: "I am tense; I am worried" and "I feel calm; I feel secure." Trait anxiety items include: "I worry too much over something that really doesn't matter" and "I am content; I am a steady person." All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety. The STAI is appropriate for those who have at least a sixth-grade reading level. Internal consistency coefficients for the scale have ranged from .86 to .95; test-retest reliability coefficients have ranged from .65 to .75 over a 2-month interval (Spielberger et al., 1983). Test-retest coefficients for this measure in the present study ranged from .69 to .89. Considerable evidence attests to the construct and concurrent validity of the scale (Spielberger, 1989).

SECONDARY OUTCOMES:
Brief Fatigue Inventory-Taiwan (BFI-T) Survey | 12 weeks
  The BFI-T scoring total ranges from0 to 90 points; a higher score corresponds to higher fatigue.
  The BFI-T's internal consistency showed a Cronbach's ! value of .97. Construct validity of the BFI-T was estimated by factor analysis with a factor loading range of 0.80 to 0.94 on a single factor. Convergent validity was examined by correlations between the BFI ''worst'' fatigue and fatigue severity scores with Profile of Mood States vigor (r = j0.69 and j0.71, respectively) and fatigue subscale scores (r = 0.82 and 0.87, respectively)(Chou, Hsieh, Yao, & Barsevick, 2016)

OTHER OUTCOMES:
WHOQOL Survey | 12 weeks
  The WHOQOL scoring total ranges from4 to20points; a higher score corresponds to good quality of life. The WHOQOL's internal consistency showed a Cronbach's value of .90. Test-retest reliability of WHOQOL was 0.75. Construct validity was examined by Person correlations (r =0.48-0.82) (Yao et al., 2000).

CONTACTS AND LOCATIONS:
Overall Officials: Chinghui Chuang, PhD, Principal Investigator — Chang Gung Medical Foundation
Locations (1):
- Chang Gung, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
we decide to share on December 2020.